CLINICAL TRIAL: NCT05827302
Title: Integrating Electronic Patient Reported Biometric Measures (ePReBMs) From the Health Gauge Phoenix Smart Watch in Respiratory Diseases
Brief Title: Integrating ePReBMs From Phoenix in Respiratory Diseases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resource Issues
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00125759
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Hypertension; COPD; Interstitial Lung Disease; Healthy Volunteers
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: The study will compare healthy controls to those with respiratory disease. Both groups will be wearing the watch and completing the same questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device: Health Gauge AI-Based Wearable Device - Model: Phoenix (Experimental)
  Interventions: Device: Health Gauge AI-Based Wearable Device - Model: Phoenix

INTERVENTIONS:
Device: Health Gauge AI-Based Wearable Device - Model: Phoenix — Wearable device

SUMMARY:
Participants with respiratory disease experience often a worsening of their condition, with increasing symptoms such as cough and shortness of breath. This worsening, often called exacerbation or flare up, impacts on the life of the participants, since they become limited in their daily activities.

Healthcare is still based today on limited times for clinical appointments to perform investigations and to meet with specialists/clinicians. Very often, these evaluations do not reflect the way the disease is limiting the patient's life.

Wearable devices offer the opportunity to collect data on physical activities and important clinical parameters (such as how the patient is active or just staying in bed during the day), on a daily basis.

The HG Phoenix AI- based Smart Watch produced by Health Gauge, an Albertan company based in Edmonton, has the potential to measure heart rate, heart rate variability, blood pressure, pulse wave velocity, respiratory rate, temperature, arterial saturation, sleep pattern (deep, light sleep, awake time), duration and time, daily physical activities (site count and distance) and calories burnt in a simple and non-invasive fashion. Ideally, these parameters could be monitored and recorded 24 hours per 7 days per week.

This study aims to demonstrate that this device can be used for a long time at home and it is comfortable to use for the participants, that it is not dangerous and, possibly, that it can help to identify exacerbations before the currently available investigations.

DETAILED DESCRIPTION:
Participants will be asked to wear the Health Gauge AI-based Wearable Device for at least 8 hours per day (ideally 24 hours), 3 days per week, for 6 months. The following data will be continuously collected from the wearable device:

heart rate, blood pressure, pulse wave velocity, respiratory rate, temperature, arterial saturation, sleep patterns, daily physical activities (step count and distance), and calories burnt.

Clinical data including demographics, radiographic, cardiac and lung functioning, diagnosis, and comorbidities will be collected from the participant's electronic medical record at baseline, 3 months, and 6 months.

Quality of life questionnaires (Saint George Respiratory Questionnaire, Medical Research Council Dyspnea Score, and EQ5-DL) will be completed by the participant through the Zamplo digital app at baseline, 3 and 6-month time points. A questionnaire on participant experience will also be administered at the 3 and 6-month time points.

Participants will be called monthly to assess patient-reported compliance with the wearable device, and adverse events (including emergency room visits and hospitalizations).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers, at least 18 years of age at the time of screening visit;
2. Fluent in English and able to follow the instructions to use the Health Gauge AI-based Wearable Device;
3. Willing and cognitively able to sign informed consent
4. Interstitial lung disease, chronic obstructive pulmonary disease, pulmonary hypertension, or a healthy control

Exclusion Criteria:

1. Pregnancy;
2. History of active (clinically significant) skin disorders;
3. History of allergic response to plastic materials;
4. Subjects with electronic implants of any kind (e.g. pacemaker);
5. Broken, damaged or irritated skin or rashes near the sensor application sites;
6. Subjects who are physically or cognitively unable to normally perform activities of daily living, assessed at the discretion of the investigator.

Exclusion Criteria for healthy control only:

1. An active medical conditions for which they are on chronic treatment with drugs;
2. Shortness of breath (any sort);
3. Chronic cough;
4. Fatigue or difficulty sleeping.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Length of time wearing device | 6 months
  Total length of time participant wears device

SECONDARY OUTCOMES:
Prediction of respiratory exacerbations- Number of emergency room visits or hospitalizations | 6 months
  Explore the possibility to predict exacerbations/flares up of the respiratory condition of the patients
Adverse Events | 6 months
  Number of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada